CLINICAL TRIAL: NCT05519891
Title: Satisfaction of 3D Printed Assistive Devices for Individuals With Physical Disabilities Living in a Long-Term Care Setting
Brief Title: 3D Printed Assistive Devices for Individuals With Physical Disabilities
Status: Completed | Type: Observational
Sponsor: Moravian University (Other)
Responsible Party: Sponsor
Other Study IDs: MoravianU: 22-0028
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Disability Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Custom 3D printed device — A 3D printed adaptation for a mobile device.

SUMMARY:
Our research aims to examine 3D printed device satisfaction when using mobile devices for individuals with physical disabilities in long-term care facilities, and the impact of the 3D printed device integration on overall occupational performance and satisfaction.

DETAILED DESCRIPTION:
This feasibility study will be conducted at Good Shepherd Rehabilitation Network (GSRN) in the collection of data examining 3D printing outcomes. The 3D printed devices are within the current normal and customary care of GSRN services, with the focus on the created 3D printed adaptations for mobile device usage (i.e. smartphone adaptations). The feasibility data will assist in understanding the satisfaction and performance of 3D printed devices for persons with a physical disability.

ELIGIBILITY:
Inclusion Criteria:

1. Being over the age of 18
2. Self-identified accessibility needs of the mobile device to address secondary to a physical accessibility limitation(s)
3. Accessibility requests of a device that has not already been addressed by 3D printing
4. Ownership or borrowing of a mobile device for personal use Operational definition of mobile devices: Mobile devices are a maximum length and width of 9.4" by 6.8" and must weigh less than 1.03 lb (e.g. dimensions of a standard iPad mini) and should be a one-handed use device with touch-screen capabilities

Exclusion Criteria:

1. Individuals with severe cognitive impairment (BIMS score of 7 or less)
2. Individuals who were unwilling to use a 3D printed device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are long-term residents of a Good Shepherd residential home, which provides 24 hour services for individuals with life-long physical disabilities, such as Cerebral Palsy, Muscular Dystrophy, Multiple Sclerosis, etc.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 3-4 weeks
  As a self-reported measure of occupational performance and occupational satisfaction, the scale ranges from 1-10, with 10 indicating a more favorable outcome in self-rated occupational performance and satisfaction.

SECONDARY OUTCOMES:
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | 3-4 weeks
  Participants will self-report satisfaction with the created and printed device and service on a Likert scale from 1-5, with 5 indicating maximum satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Benham, OTD, Principal Investigator — Moravian University
Locations (1):
- Moravian University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mao HF, Chen WY, Yao G, Huang SL, Lin CC, Huang WN. Cross-cultural adaptation and validation of the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0): the development of the Taiwanese version. Clin Rehabil. 2010 May;24(5):412-21. doi: 10.1177/0269215509347438. PMID 20442253
- [Background] Chodosh J, Edelen MO, Buchanan JL, Yosef JA, Ouslander JG, Berlowitz DR, Streim JE, Saliba D. Nursing home assessment of cognitive impairment: development and testing of a brief instrument of mental status. J Am Geriatr Soc. 2008 Nov;56(11):2069-75. doi: 10.1111/j.1532-5415.2008.01944.x. PMID 19016941
- [Background] Law, M., Baptiste, S., Carswell, A., McColl, M. A., Polatajko, H., & Pollock, N. (2014). Canadian Occupational Performance Measure (5th ed.). Ottawa: CAOT Publications.